CLINICAL TRIAL: NCT00271791
Title: Prednisone Treatment for Vestibular Neuronitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Collaborators: Clalit Health Services, Haifa and West Galilee (Other); Hillel Yaffe Medical Center (Other Government); Rambam Health Care Campus (Other); University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 42352; 20050277
Record Dates: First submitted 2006-01-01; First posted 2006-01-04 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-07

CONDITIONS: Vestibular Diseases; Vestibular Neuronitis
Keywords: Vestibular Neuronitis; Vestibular Function Tests; Vestibular Adaptation; Steroids
MeSH Terms: conditions — Vestibular Diseases; Vestibular Neuronitis | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Prednisone
  Interventions: Drug: Prednisone
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — PO, 1 mg/kg body weight, 5 days Short tapering regimen: daily reductions in the dose, 12 days
  Arms: 1
Drug: Prednisone — PO, Placebo, 17 days
  Arms: 2

SUMMARY:
The purpose of the study is to investigate the value of steroids in the treatment of vestibular neuronitis. The potential benefits of steroid therapy would be analyzed by the clinical response, self-perceived handicap and laboratory parameters.

DETAILED DESCRIPTION:
Vestibular neuronitis is the second most common cause of peripheral vestibulopathy (the first being benign paroxysmal positional vertigo) with incidence of about 3.5/100000. Currently vestibular neuronitis is explained by a viral pathogenesis.

Vestibular neuronitis is considered to have a benign course. The static rotatory vertigo and disequilibrium, present even when the patient is completely at rest, subside in most cases within a few days, and a gradual return to daily activities is the rule. However, it has been shown that there is generally incomplete restoration of peripheral function, and clinical recovery is achieved by proprioceptive and visual substitution for the unilateral vestibular deficit, combined with central vestibular compensation of the imbalance in vestibular tone. Although vestibular neuronitis is usually restricted to one attack, several studies have reported continuous or episodic vertigo or unsteadiness in 43% -53% of patients. The main residua include impaired vision and disequilibrium during walking and especially during head movement toward the affected ear. The rate of positive finding on vestibular evaluation may reach 60%. However, vestibular impairment as reflected by positive bedside testing and vestibular laboratory evaluation is not necessarily accompanied by subjective complaints and does not always reflect the level of incapacity.

The assumed HSV-1 etiology of vestibular neuronitis and the reported benefit of the combination of steroids and acyclovir in Bell's palsy suggest similar advantage in the treatment of vestibular neuronitis. Also, glucocorticoid receptors activation was reported to enhance vestibular compensation after acute peripheral vestibular insults in various animal models. A recent study investigated the effect of prednisolone versus valacyclovir and placebo on canal paresis in vestibular neuronitis patients. It was found that steroid treatment significantly improved peripheral vestibular function to the extent reflected by the caloric testing. However, bedside findings, patients' complaints and daily handicap were not evaluated. The relevance of the EOG caloric test results to clinical improvement could be argued in light of a previous report showing no correlation between EOG findings and residual symptoms in a long-term follow-up of vestibular neuronitis patients, and the finding that corticosteroid therapy had no effect on symptoms despite significant recovery of the caloric-test results.

The purpose of the study:

Prospective controlled longitudinal 12-month evaluation of the value of steroids in the treatment of vestibular neuronitis. The potential benefits of steroid therapy would be analyzed by the clinical response, self-perceived handicap and EOG laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of vestibular neuronitis.
* Documentation of unilateral reduced caloric response (caloric asymmetry >25%) on the EOG caloric study.

Exclusion Criteria:

* Complaints of new hearing loss, tinnitus, or neurological deficits.
* The presence of previously non-diagnosed sensorineural hearing loss (SNHL)
* History of vestibular dysfunction.
* Patient younger than 18 years of age.
* Known contra-indication to systemic steroids: Unbalanced hypertension, un-controlled diabetes mellitus, immunodeficiency, active peptic disease, and avascular necrosis of the femoral head.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-09; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Clinical: The presence of static and dynamic nystagmus, positional and positioning nystagmus, and disequilibrium on bedside examination. | 12 months

SECONDARY OUTCOMES:
Functional: Scores on the Dizziness Handicap Inventory questionnaires. | 12 months
Laboratory: Caloric lateralization and directional preponderance on electro-oculography (EOG). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Avi Shupak, MD, Principal Investigator — Carmel Medical Center and Clalit Health Services, Haifa and West Galilee; Itzhak Braverman, MD, Principal Investigator — Hillel Yaffe Medical Center; Avishai Golz, MD, Principal Investigator — Rambam Health Care Campus; Elhanan Greenberg, ND, Principal Investigator — Carmel Medical Center; Avi Shupak, MD, Study Chair — Carmel Medical Center and Clalit Health Services, Haifa and West Galilee
Locations (4):
- Israel (4):
  - Unit of Otolaryngology Head and Neck Surgery, Hillel Yaffe Medical Center, Hadera
  - Department of Otolaryngology Head and Neck Surgery, Rambam Medical Center, Haifa
  - Department of Otolaryngology Head and Neck Surgery, Carmel Medical Center, Haifa
  - Otoneurolgy Unit, Lin Medical Center, Clalit Health Services, Haifa

REFERENCES:
- [Background] Strupp M, Zingler VC, Arbusow V, Niklas D, Maag KP, Dieterich M, Bense S, Theil D, Jahn K, Brandt T. Methylprednisolone, valacyclovir, or the combination for vestibular neuritis. N Engl J Med. 2004 Jul 22;351(4):354-61. doi: 10.1056/NEJMoa033280. PMID 15269315
- [Background] Ohbayashi S, Oda M, Yamamoto M, Urano M, Harada K, Horikoshi H, Orihara H, Kitsuda C. Recovery of the vestibular function after vestibular neuronitis. Acta Otolaryngol Suppl. 1993;503:31-4. doi: 10.3109/00016489309128067. PMID 8470496
- [Background] Ariyasu L, Byl FM, Sprague MS, Adour KK. The beneficial effect of methylprednisolone in acute vestibular vertigo. Arch Otolaryngol Head Neck Surg. 1990 Jun;116(6):700-3. doi: 10.1001/archotol.1990.01870060058010. PMID 2187486
- [Background] Arbusow V, Schulz P, Strupp M, Dieterich M, von Reinhardstoettner A, Rauch E, Brandt T. Distribution of herpes simplex virus type 1 in human geniculate and vestibular ganglia: implications for vestibular neuritis. Ann Neurol. 1999 Sep;46(3):416-9. doi: 10.1002/1531-8249(199909)46:33.0.co;2-w. PMID 10482275
- [Background] Bergenius J, Perols O. Vestibular neuritis: a follow-up study. Acta Otolaryngol. 1999;119(8):895-9. doi: 10.1080/00016489950180243. PMID 10728930
- [Background] Shupak A, Nachum Z, Stern Y, Tal D, Gil A, Gordon CR. Vestibular neuronitis in pilots: follow-up results and implications for flight safety. Laryngoscope. 2003 Feb;113(2):316-21. doi: 10.1097/00005537-200302000-00022. PMID 12567089
- [Background] Cameron SA, Dutia MB. Lesion-induced plasticity in rat vestibular nucleus neurones dependent on glucocorticoid receptor activation. J Physiol. 1999 Jul 1;518(Pt 1):151-8. doi: 10.1111/j.1469-7793.1999.0151r.x. PMID 10373697
- [Background] Fife TD, Tusa RJ, Furman JM, Zee DS, Frohman E, Baloh RW, Hain T, Goebel J, Demer J, Eviatar L. Assessment: vestibular testing techniques in adults and children [RETIRED]: report of the Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology. Neurology. 2000 Nov 28;55(10):1431-41. doi: 10.1212/wnl.55.10.1431. No abstract available. PMID 11094095